CLINICAL TRIAL: NCT06345742
Title: The Effect of Parental Participation on Newborn Comfort During Diaper Care Practice in Preterm Infants
Brief Title: The Effect of Parental Participation on Newborn Comfort During Diaper Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Zehra Kan Onturk, Assist. Prof., Acibadem University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ATADEK-2023-10/396
Record Dates: First submitted 2024-03-26; First posted 2024-04-03 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-03

CONDITIONS: Preterm
Keywords: diaper care; newborn comfort; parental participation; preterm
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control group (no parental participation) (Other): In the control group, infant diaper care will be carried out without parental participation.
  Interventions: Other: No parental participation
- Experimental group (mother participation) (Experimental): In the experimental group, infant diaper care will be provided with the mothers.
  Interventions: Other: Mother participation
- Experimental group (father participation) (Experimental): In the experimental group, infant diaper care will be provided with the fathers.
  Interventions: Other: Father participation

INTERVENTIONS:
Other: No parental participation — 1. Before collecting data, Preterm Infant information form will be filled out.
  2. The "Premature Infant Comfort Scale" will be evaluated before the procedure.
  3. Diaper care will be performed by the primary nurse.
  4. "Premature Infant Comfort Scale" will be evaluated during and after the diaper care application.
  Arms: Control group (no parental participation)
Other: Mother participation — 1. Before collecting data, Preterm Infant information form will be filled out.
  2. The "Premature Infant Comfort Scale" will be evaluated before the procedure.
  3. Mothers' stress level will be determined using the "Neonatal Intensive Care Unit Parent Stress Scale"
  4. Mothers will be given practical diaper care training on the infant model doll.
  5. Diaper care will be provided by the mothers of the infants
  6. "Premature Infant Comfort Scale" will be evaluated during and after the application.
  Arms: Experimental group (mother participation)
Other: Father participation — 1. Before collecting data, Preterm Infant information form will be filled out.
  2. The "Premature Infant Comfort Scale" will be evaluated before the procedure.
  3. Fathers' stress level will be determined using the "Neonatal Intensive Care Unit Parent Stress Scale"
  4. Fathers will be given practical diaper care training on the infant model doll.
  5. Diaper care will be provided by the fathers of the infants
  6. "Premature Infant Comfort Scale" will be evaluated during and after the application.
  Arms: Experimental group (father participation)

SUMMARY:
It was aimed to determine the effect of parental participation on newborn comfort during diaper care practice in preterm infants.

H1: Parental participation during infant diaper care practice in preterm infants has an effect on newborn comfort.

H2: There is a difference in the effect of parent diaper care practice and the participation of the mother or father on newborn comfort in preterm infants.

H3: There is a difference between the stress levels of parents before the application of infant diaper care in preterm infants.

DETAILED DESCRIPTION:
The expectation of all parents is to have a healthy baby at the end of the pregnancy. However, newborns being born unexpectedly early and being admitted to the neonatal intensive care unit is a stressful situation for both newborns and parents. During this process, parents of preterm infants experience anxiety, loss of control, fear of the future, depression, role change and concerns about the improvement of the baby's condition. It is important for parents to actively participate in care within the framework of family-centered care practices in order to reduce the newborn's stress level, increase its comfort and improve its environment and to increase the families' ability to cope with this situation.Infant care, which is repeated many times a day in the Neonatal Intensive Care Unit, is one of the care practices that include tactile stimuli. Studies have observed that preterm infants' stress increases during diaper changes. For this reason, it is important to plan the necessary invasive practices to increase comfort during diaper changes, to include parental participation in these procedures, and to determine the effect of these interventions on the infants' comfort and to include them in the literature.

ELIGIBILITY:
Inclusion Criteria:

* Infants whose gestational age is between ≥34 weeks and ≤36+6 weeks at the time of application
* Infants with stable health conditions

Exclusion Criteria:

* Intubated
* Those with very low and extremely low birth weight at the time of procedure
* Having a chronic disease
* Those with congenital anomalies
* Having undergone a surgical procedure
* Having neurological symptoms
* Receiving oxygen support
* Diagnosed with sepsis
* Sedated
* A pharmacological analgesic method was used four hours before.
* Parents who do not want to participate in care

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 105 (Actual)
Dates: Start 2023-12-19 (Actual); Primary Completion 2024-10-18 (Actual); Study Completion 2024-10-18 (Actual)

PRIMARY OUTCOMES:
Level of Parental Stress | It will be measured once just before the diaper care
  The level of parental stress will be measured using the Neonatal Intensive Care Unit Parental Stress Scale.The scale was developed by Miles, Funk and Carlson in 1993 to determine the perception levels of stressors arising from the physical and psychosocial environment by mothers and fathers. The Turkish validity and reliability study of the scale was conducted by Turan and Başbakkal in 2006. The scale consists of 5 rating points and is rated from 1 (not stressful) to 5 (extremely stressful). The score that can be obtained from the scale varies between 0 and 170. The scale can be applied to mothers and fathers with infants in the neonatal intensive care unit
Change in Level of Comfort | immediately before the procedure, during the procedure, immediately after the procedure. The change in these time intervals will be assessed
  The infants' comfort level will be measured using the Premature Infant Comfort Scale.The scale is a multi-dimensional scale used to measure comfort in preterm newborns. The Premature Infant Comfort Scale was developed by Monique et al. in the Netherlands in 2007. The validity and reliability of the Turkish scale was determined by Küçük Alemdar and Güdücü Tüfekçi in 2015. The scale consists of 1 to 5 rating points. The infant's comfort is evaluated based on the total score according to the scale. According to the total score, 35 indicates the lowest score, 7 indicates the highest comfort level, and a high score indicates a low comfort level. The subscales of the scale include the preterm infant's alertness, calmness, respiratory status, physical movement, muscle tone, facial movements, and average heart rate

CONTACTS AND LOCATIONS:
Overall Officials: Tuğba Turker, Nurse, Principal Investigator — Acibadem University
Locations (1):
- Acıbadem University, Istanbul, Ataşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Girabent-Farres M, Jimenez-Gonzalez A, Romero-Galisteo RP, Amor-Barbosa M, Bagur-Calafat C. Effects of early intervention on parenting stress after preterm birth: A meta-analysis. Child Care Health Dev. 2021 May;47(3):400-410. doi: 10.1111/cch.12853. Epub 2021 Feb 15. PMID 33559337
- [Background] Miles MS, Funk SG, Carlson J. Parental Stressor Scale: neonatal intensive care unit. Nurs Res. 1993 May-Jun;42(3):148-52. PMID 8506163
- [Background] Morelius E, Hellstrom-Westas L, Carlen C, Norman E, Nelson N. Is a nappy change stressful to neonates? Early Hum Dev. 2006 Oct;82(10):669-76. doi: 10.1016/j.earlhumdev.2005.12.013. Epub 2006 Feb 28. PMID 16507341
- [Background] Pichler-Stachl E, Urlesberger P, Mattersberger C, Baik-Schneditz N, Schwaberger B, Urlesberger B, Pichler G. Parental Stress Experience and Age of Mothers and Fathers After Preterm Birth and Admission of Their Neonate to Neonatal Intensive Care Unit; A Prospective Observational Pilot Study. Front Pediatr. 2019 Oct 24;7:439. doi: 10.3389/fped.2019.00439. eCollection 2019. PMID 31709208
- [Background] Prouhet PM, Gregory MR, Russell CL, Yaeger LH. Fathers' Stress in the Neonatal Intensive Care Unit: A Systematic Review. Adv Neonatal Care. 2018 Apr;18(2):105-120. doi: 10.1097/ANC.0000000000000472. PMID 29595549